CLINICAL TRIAL: NCT02540018
Title: Multicenter Randomized Controlled Trial to Assess the Effectiveness of Paclitaxel-coated Luminor® Balloon Catheter Versus Uncoated Balloon Catheter in the Superficial Femoral and Popliteal Arteries to Prevent Vessel Restenosis or Reocclusion
Brief Title: Effectiveness of Paclitaxel-coated Luminor® Balloon Catheter Versus Uncoated Balloon Catheter in the Arteria Femoralis Superficialis
Acronym: EffPac
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jena University Hospital (Other)
Collaborators: iVascular S.L.U. (Industry); KKS Netzwerk (Network)
Responsible Party: Principal Investigator, Ulf Teichgräber, Principal Investigator, Jena University Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CIV-15-03-013204
Record Dates: First submitted 2015-08-17; First posted 2015-09-03 (Estimated); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Peripheral Arterial Disease
Keywords: DEB, drug-eluting balloon, Paclitaxel, peripheral artery disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Angioplasty; Catheters

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paclitaxel-coated Luminor® Balloon Catheter (Active Comparator): The balloon dilatation procedure, including deployment to the target lesion and balloon inflation, deflation and retrieval, is performed under fluoroscopic observation. An endoluminal guidewire passage of the stenotic and occlusive femoro-popliteal lesion is mandatory. After pre-dilatation of the target lesion an angiographic assessment will be performed (DSA or XA). Randomization will be performed by envelope pull. The treatment group represents the Luminor® DEB PTA. After dilation of the target lesion, the PTA catheter is withdrawn through the introducer sheath, and a post-PTA angiography is performed (DSA or XA) to evaluate the technical result and possible procedural complications. A final run-off angiography (DSA or XA) of the BTK arteries is required.
  Interventions: Device: Transluminal Angioplasty with Paclitaxel-coated Luminor® Balloon Catheter in the Superficial Femoral and Popliteal Arteries
- Uncoated Balloon Catheter (Active Comparator): Identical procedure also for control arm with PTA balloon (see below): After pre-dilatation, randomization will be performed by envelope pull. The control group requires an uncoated balloon catheter. After dilation of the target lesion, the PTA catheter is withdrawn and a post-PTA angiography is performed (DSA or XA) to evaluate the technical result and possible procedural complications. A final run-off angiography (DSA or XA) of the BTK arteries is required.
  Interventions: Device: Transluminal Angioplasty with and non-coated (CE-marked) plain old angioplasty balloon (POBA) catheter

INTERVENTIONS:
Device: Transluminal Angioplasty with Paclitaxel-coated Luminor® Balloon Catheter in the Superficial Femoral and Popliteal Arteries — Endoluminal guidewire passage of the stenotic and occlusive femoro-popliteal lesion must be performed. A pre-dilatation follows. Then the investigational procedure (DEB) is assigned by randomization.
  Luminor35®-DEB PTA catheter is applied.
  Other Names: DEB
  Arms: Paclitaxel-coated Luminor® Balloon Catheter
Device: Transluminal Angioplasty with and non-coated (CE-marked) plain old angioplasty balloon (POBA) catheter — Endoluminal guidewire passage of the stenotic and occlusive femoro-popliteal lesion must be performed. A pre-dilatation follows. Then the investigational procedure is assigned by randomization. POBA catheter is applied.
  Other Names: POBA
  Arms: Uncoated Balloon Catheter

SUMMARY:
The aim of this clinical trial is to evaluate the safety and efficacy of the novel Luminor® paclitaxel drug-eluting balloon (iVascular, S.L.U., Barcelona, Spain) in inhibiting restenosis and in ensuring long-term patency.

DETAILED DESCRIPTION:
The investigational medical device represents the Paclitaxel drug-eluting Luminor®-35 balloon catheter which is based on a proprietary transfertech coating technology. This has been engineered to improve clinical efficacy by optimizing coating properties and device functionalities. This allows a homogeneous and precise Paclitaxel concentration of 3 μg/mm2 on the PTA balloon surface. The balloon dilatation procedure, including deployment to the target lesion and balloon inflation, deflation and retrieval, is performed under fluoroscopic observation. All sites shall have access to an emergency unit to perform also interventions as bypass surgery e.g. in case of failed percutaneous transluminal angioplasty (PTA). The patient is positioned on the angiographic table and draped in a sterile fashion. The standard vascular access represents the ipsilateral or contralateral femoral artery in accordance to the target vessel. The endovascular procedure can be performed in a direct antegrade or a cross-over retrograde technique.

An introducer sheath will be inserted over a guidewire. 5.000 I.U. heparin is injected i.a. to pre-vent peri-procedural thrombotic events. Alternative peri-procedural anti-coagulation regimens may be applied if justified by individual patient requirements. An endoluminal guidewire passage of the stenotic and occlusive femoro-popliteal lesion is mandatory for study inclusion.

A POBA PTA balloon of appropriate balloon diameter and length, and catheter working length is selected according to the characteristics of the target vessel and lesion for the pre-dilation and assessed by angiography (DSA or XA). A ruler has to be adjacent to the target vessel. After pre-dilatation of the target lesion an angiographic assessment will be performed (DSA or XA). A ruler has to be adjacent to the target vessel.

Randomization will be performed by envelope pull. The treatment group represents the Lumi-nor® DEB and the control group POBA applying a CE-marked non-drug-eluting PTA balloon catheter. In patients with peripheral artery disease, quantitative vascular angiography (QVA) is essential for the analysis of the degree of the arterial stenosis. For quantitative assessment of stenotic lesions, the residual lumen at the lesion site is compared with the lumen at a reference site.

QVA will be assessed by an independent core lab. The assessment during the angioplasty is performed pre- and post-procedure, at 6 months follow-up and any unscheduled procedure if necessary. Follow-up (FU) assessments will occur at pre-discharge, 6, 12 and 24 months following the study procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Subject must agree to undergo the 6-month angiographic and clinical follow-up (at 12 month post-procedure)
3. Peripheral vascular disease Rutherford class 2-4
4. De novo stenotic/re-stenotic lesion or occlusive lesions in the superficial femoral (SFA) and/or popliteal arteries (PA)
5. If the index lesion is re-stenotic, the prior PTA must have been >30 days prior to treatment in the current study
6. ≥70% diameter stenosis or occlusion
7. Target lesion length: ≤15 cm (TASC II A and B)
8. Only one lesion per limb and per patient can be treated (see definition chapter 6.5)
9. ≥ one patent intrapopliteal run-off artery to the foot of the index limb
10. Successful endoluminal guidewire passage through the target lesion
11. Predilatation prior to randomization
12. Life expectancy, in the investigators opinion of at least one year
13. Subject is able to verbally acknowledge and understand the aim of this trial and is willing and able to provide informed consent

Exclusion Criteria:

1. Previous surgery in the target vessel
2. Major amputation in the same limb as the target lesion
3. Presence of aneurysm in the target vessel
4. Acute myocardial infarction within 30 days before intervention
5. Severely calcified target lesions in the SFA/PA resistant to PTA
6. Subjects requiring different treatment or raising serious safety concern regarding the procedure or the required medication
7. Women of childbearing potential expect women with the following criteria:

   * post-menopausal (12 month natural amenorrhea or 6 month amenorrhea with serum FSH > 40mlU/ml)
   * sterilization 86 weeks after bilateral ovariectomy with or without hysterectomy
   * using an effective method of birth control for the duration of the trial: implants, injectables, combined oral contraceptives, intrauterine device (in place for a period of at least 2 months prior to screening) and with negative serum pregnancy test
   * sexual abstinence
   * vasectomy partner
8. Pregnant and nursing women
9. Acute thrombus, stent or aneurysm in the index limb or vessel
10. Renal insufficiency with a serum creatinine >2.0 mg/dL at baseline
11. Platelet count <50 G/l or >600 G/l at baseline
12. Known hypersensitivity or contraindication to contrast agent that cannot be adequately pre-medicated
13. Subjects with known allergies against Paclitaxel
14. Subjects with intolerance to antiplatelet, anticoagulant, or thrombolytic medications that would be administered during the trial
15. Dialysis or immunosuppressant therapy
16. Current participation (or within the last 3 months) in another interventional study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2015-09-15 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Change in Late Lumen Loss (LLL) | at baseline and after 6 months
  Change in Late Lumen Loss (LLL), defined as difference between the diameters (in mm) at 6 months follow-up minus post-procedure.

SECONDARY OUTCOMES:
Revascularisation of TVR | after 6 months and 12 months
  Freedom of target vessel revascularization (TVR)
Revascularisation of TLR | after 6 months and 12 months
  Freedom from target lesion revascularization (TLR)
Change in Rutherford classification | after 6 months and 12 months
  Change of Rutherford stage to baseline at Follow-up
Change of ABI | after 6 months and 12 months
  Decrease in the ankle-brachial-index
Change of Life Quality | after 6 months and 12 months
  Improvement of life quality according to the Walking Impairment Questionnaire (WIQ) and the EQ5D questionnaire to baseline at Follow-up
Absence of amputation | after 6 months and 12 months
  Major and minor amputation rate at the index limb
Bailouts | after 6 months and 12 months
  Number of bailouts
Mortality | after 6 months and 12 months
  Mortality rate independently of the direct cause

CONTACTS AND LOCATIONS:
Overall Officials: René Aschenbach, PD Dr. med., Principal Investigator — University Hospital Jena, Radiology
Locations (11):
- Germany (11):
  - Herzzentrum Bad Krozingen, Bad Krozingen, Baden-Wurttemberg
  - SRH Klinikum Karlsbad-Langensteinbach, Karlsbad-Langensteinbach, Baden-Wurttemberg
  - Institut für Klinische Radiologie, Klinikum der Ludwig Maximilians Universität München - Campus Innenstadt, München, Bavaria
  - Westpfalz-Klinikum GmbH Standort II Kusel, Kusel, Rhineland-Palatinate
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Klinikum Arnsberg Angiologie, Arnsberg, Thuringia
  - University Hospital Jena, Radiology, Jena, Thuringia
  - Medinos Kliniken Sonneberg, Sonneberg, Thuringia
  - Ihre-Radiologen Berlin Gemeinschaftspraxis für Radiologie, Berlin
  - Angiologikum Hamburg, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg

REFERENCES:
- [Derived] Teichgraber U, Lehmann T, Ingwersen M, Aschenbach R, Zeller T, Brechtel K, Blessing E, Lichtenberg M, von Flotow P, Heilmeier B, Sixt S, Brucks S, Erbel C, Beschorner U, Werk M, Riambau V, Wienke A, Klumb C, Thieme M, Scheinert D. Long-Term Effectiveness and Safety of Femoropopliteal Drug-Coated Balloon Angioplasty : 5-Year Results of the Randomized Controlled EffPac Trial. Cardiovasc Intervent Radiol. 2022 Dec;45(12):1774-1783. doi: 10.1007/s00270-022-03265-1. Epub 2022 Sep 11. PMID 36088609
- [Derived] Teichgraber U, Lehmann T, Aschenbach R, Scheinert D, Zeller T, Brechtel K, Blessing E, Lichtenberg M, Sixt S, Brucks S, Beschorner U, Klumb CT, Thieme M; Collaborators. Efficacy and safety of a novel paclitaxel-nano-coated balloon for femoropopliteal angioplasty: one-year results of the EffPac trial. EuroIntervention. 2020 Apr 3;15(18):e1633-e1640. doi: 10.4244/EIJ-D-19-00292. PMID 31687933
- [Derived] Teichgraber U, Aschenbach R, Scheinert D, Zeller T, Brechtel K, Thieme M, Blessing E, Treitl M, Lichtenberg M, von Flotow P, Vogel B, Werk M, Riambau V, Wienke A, Lehmann T, Sixt S. The effectiveness of the paclitaxel-coated Luminor(R) balloon catheter versus an uncoated balloon catheter in superficial femoral and popliteal arteries in preventing vessel restenosis or reocclusion: study protocol for a randomized controlled trial. Trials. 2016 Oct 28;17(1):528. doi: 10.1186/s13063-016-1657-x. PMID 27793175